CLINICAL TRIAL: NCT01759394
Title: A Randomized, Open-label, Three-period, Partial-replicate Design Study to Evaluate the Inter- and Intrasubject Variability of the Avatrombopag To-be-marketed Formulation Administered as Single Doses of 40 mg to Healthy Subjects Receiving a Low-fat Meal
Brief Title: A Open-label, Three-period, Partial-replicate Design Study to Evaluate the Inter- and Intrasubject Variability of the Avatrombopag To-be-marketed Formulation Administered as Single Doses of 40 mg to Healthy Subjects Receiving a Low-fat Meal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E5501-A001-017
Record Dates: First submitted 2012-12-06; First posted 2013-01-03 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — avatrombopag

ARMS (1):
- Avatrombopag maleate 40 mg (Experimental)
  Interventions: Drug: Avatrombopag maleate 40 mg

INTERVENTIONS:
Drug: Avatrombopag maleate 40 mg — Avatrombopag maleate 40 mg (2 x 20 mg tablets- all doses are expressed as avatrombopag, the amount of free base) given with 240 mL water in three single oral doses, one during each of three treatment periods. Participants randomized to one of three treatment sequences:
  * Fed, Fed, Fasted; or
  * Fed, Fasted, Fed; or
  * Fasted, Fed, Fed
  During the Fasted period, participants must have fasted for at least a 10-hour overnight fast and to refrain from eating for 4 hours.
  During the Fed period, participants were allowed approximately 30 minutes to eat a low-fat breakfast and required to take the drug within 15 minutes of completion of breakfast.
  Randomization Phase consists of three single-dose treatment periods:
  Treatment Period 1 and 2 separated by a 7-day washout interval. Treatment Period 2 and 3 separated by a 28-day washout interval. Treatment period 3 and the Follow-up/ Termination Visit will be separated by a 30-day (+1 day) washout interval.
  Other Names: E5501

SUMMARY:
A Randomized, Open-label, Three-period, Partial-replicate Design Study to Evaluate the Inter- and Intrasubject variability of the Avatrombopag To-be-marketed Formulation Administered as Single Doses of 40 mg (all doses are expressed as avatrombopag, the amount of free base) to healthy subjects Receiving a low-fat Meal.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study:

1. Healthy male and female subjects (aged 18 to 55 years inclusive, at the time of informed consent)
2. Body mass index (BMI) ≥ 18 kg/m2 and ≤ 32 kg/m2 at Screening
3. Platelet count between 120 x 109/L and 300 x 109/L inclusive at Screening, Baseline Period 1, or Baseline Period 3
4. Platelet count below the upper limit of normal at Baseline Period 2
5. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative serum beta-human chorionic gonadotropin [β-hCG] test with a minimum sensitivity 25 IU/L or equivalent units of β-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
6. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
7. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, a nonhormonal-based intrauterine device, a double barrier method [such as condom plus spermicide or diaphragm plus spermicide], non-estrogen-based hormonal therapy, progesterone-only contraceptive implant/injection, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the subject must agree to use a double barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. The use of estrogen-based hormonal contraceptives is not allowed because of a potential increase in the risk of venous thrombosis.

   All females who are of reproductive potential and have been using estrogen-containing oral contraceptives must have discontinued the contraceptive product for at least 30 days before dosing, throughout the entire study period, and for 30 days after study drug discontinuation, and have been using use the aforementioned methods.
8. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 90 days after study drug discontinuation). No sperm donation is allowed during the study period and for at least 90 days after the last dose of study drug.
9. Provide written informed consent
10. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Evidence of clinically significant cardiovascular, hepatic, gastrointestinal, renal, respiratory, endocrine, hematologic, neurologic, or psychiatric disease or abnormalities or a known history of any gastrointestinal surgery that could impact the PK of study drug
2. Agents associated with thrombotic events (including oral contraceptives) are required to be discontinued 30 days prior to first study drug administration
3. Evidence of organ dysfunction or any clinically significant deviation from normal in medical history, e.g., history of splenectomy
4. History of arterial or venous thrombosis, including partial or complete thromboses (e.g., stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, or pulmonary embolism)
5. Known family history of hereditary thrombophilic disorders (e.g., Factor V Leiden, antithrombin III deficiency, etc.)
6. Hemoglobin less than the lower limit of normal
7. Clinically significant illness within 8 weeks, or a clinically significant infection within 4 weeks, of dosing
8. Evidence of clinically significant deviation from normal in physical examination, vital signs, or clinical laboratory determinations at Screening or Baseline Periods 1 or 3
9. A corrected QT interval using Fridericia's formula (QTcF) > 450 ms at Screening
10. A known or suspected history of drug or alcohol misuse within 6 months before Screening, or a positive drug test at Screening or Baseline Periods 1 or 3
11. Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), and hepatitis C antibody (HCVAb) tests at Screening
12. Receipt of blood products within 4 weeks, donation of blood within 8 weeks, or donation of plasma within 1 week before dosing
13. Known history of clinically significant drug or food allergies or experiencing significant seasonal allergy (e.g., hay fever) or hypersensitivity to avatrombopag and/or any of its excipients
14. Use of prescription drugs within 4 weeks or within five times the drug's half-life (if that time is >4 weeks) before Screening
15. Participation in another clinical trial within 60 days before dosing or concurrent enrollment in another clinical trial
16. Unwilling or unable to abide by the requirements of the study
17. Any condition that would make them, in the opinion of the investigator, unsuitable for the study or who, in the opinion of the investigator, are not likely to complete the study for any reason
18. Females who are pregnant (positive β-hCG test) or breastfeeding
19. Hypersensitivity to aspirin
20. Scheduled for surgery or other invasive procedure during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time course profile From Time = 0 to time extrapolated to infinity (AUC [0-inf]) | predose (-60 minutes), 1, 2, 3, 4, 5, 6, 7, 8, 12, 18, 24, 36, 48, 72, and 96 hours postdose
  AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Maximum Observed Plasma Concentration (Cmax) | predose (-60 minutes), 1, 2, 3, 4, 5, 6, 7, 8, 12, 18, 24, 36, 48, 72, and 96 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Mark Allison, MD, Principal Investigator — Eisai Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States